CLINICAL TRIAL: NCT06571344
Title: Vitamin D in Dialysis Patients - Diagnostic and Therapeutic Management
Status: Recruiting | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: NKBBN/783/2022
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Vitamin D Deficiency Due to Chronic Kidney Disease
Keywords: vitamin D; cholecalciferol; 25-hydroxycholecalciferol; parathyroid hormone; FGF23; GDF15; chronic kidney disease-mineral and bone disorder; dialysis
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Cholecalciferol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 25(OH)D < 30 ng/mL: Dialysed patients with vitamin D level (25(OH)D) < 30 ng/mL administered cholecalciferol
  Interventions: Drug: Cholecalciferol
- 25(OH)D 30 - 49.9 ng/mL: Dialysed patients with vitamin D level (25(OH)D) 30-49.9 ng/mL administered cholecalciferol
  Interventions: Drug: Cholecalciferol
- 25(OH)D 50-80 ng/mL: Dialysed patients with vitamin D level (25(OH)D) 50-80 ng/mL administered cholecalciferol
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — The patients with vitamin D (25(OH)D) levels < 30 ng/mL, and 30-50 ng/ml will recieve a dose of cholecalciferol at 70,000 IU per week (20,000 IU + 20,000 IU + 30,000 IU per week).
  In the patients with 25(OH)D levels 50-80 ng/mL the dose of cholecalciferol will be adjusted to avoid exceeding the upper limit of the laboratory norm.

SUMMARY:
The goal of this observational study is to learn about the effects of cholecalciferol administration, according to guidelines for the general population, on laboratory parameters of Chronic Kidney Disease-Mineral and Bone Disorder in dialysis patients, depending of the attained levels of vitamin D (25OH)D).

The main question it aims to answer is:

How does cholecalciferol affect calcium and phosphate metabolism parameters depending on the achieved levels of 25(OH)D?

Participants taking cholecalciferol as part of their regular medical care for CKD-MBD will have the laboratory result parameters observed for up to 4 years.

DETAILED DESCRIPTION:
The analysis will involve data obtained from medical records of dialysis patients who receive standard procedures consistent with national and international guidelines for specialized care.

Specifically, we will analyze the levels of:

* 25(OH)D,
* 1,25(OH)2D
* Calcium
* Phosphates
* PTH
* FGF23
* GDF15 to assess the efficacy and safety of cholecalciferol in dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 5,dialysed patients with vitamin D deficiency or insufficiency (level of 25(OH)D < 30 ng/mL)

Exclusion Criteria:

* dialysis time of less than 3 months
* inadequately controled secondary hyperparathyroidism (iPTH>800pg/mL)
* treatment with calcimimetics
* treatment with active forms of vitamin D3,
* parathyroidectomy
* bilateral nephrectomy
* treatment with corticosteroids
* lack of consent to take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in Department of Nephrology Transplantology and Internal Medicine, Medical University of Gdansk
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
efficacy and safety of cholecalciferol therapy in dialysed patients | 2022-2026
  analysis of - vitamin D levels - 25(OH)D, 1,25(OH)2D, calcium-phosphate metabolism parameters (serum calcium, phosphate, PTH levels),FGF23, GDF15 levels, in 3 groups of patients achieving different range of 25(OH)D levels

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Tylicki, Prof., Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdansk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pludowski P, Takacs I, Boyanov M, Belaya Z, Diaconu CC, Mokhort T, Zherdova N, Rasa I, Payer J, Pilz S. Clinical Practice in the Prevention, Diagnosis and Treatment of Vitamin D Deficiency: A Central and Eastern European Expert Consensus Statement. Nutrients. 2022 Apr 2;14(7):1483. doi: 10.3390/nu14071483. PMID 35406098
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD-MBD Update Work Group. KDIGO 2017 Clinical Practice Guideline Update for the Diagnosis, Evaluation, Prevention, and Treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD). Kidney Int Suppl (2011). 2017 Jul;7(1):1-59. doi: 10.1016/j.kisu.2017.04.001. Epub 2017 Jun 21. No abstract available. PMID 30675420